CLINICAL TRIAL: NCT05417737
Title: Prospective and Observational Study of Patients Referred to the Chronic Pain Unit for Palliative Treatment With Ozone Therapy Between 2022 and 2025. (EPOOzo)
Brief Title: Patients Referred to the Chronic Pain Unit for Palliative Treatment With Ozone Therapy Between 2022 and 2025
Acronym: EPOOzo
Status: Recruiting | Type: Observational
Sponsor: Bernardino Clavo, MD, PhD (Other)
Collaborators: Fundacion Canaria Instituto de Investigacion Sanitaria de Canarias (Other); Servicio Canario de Salud (Other); Council of Gran Canaria (Other); Red de Investigación en Servicios de Salud en Enfermedades Crónicas (Other); Instituto Universitario de Enfermedades Tropicales y Salud Pública de Canarias, Universidad de La Laguna (Unknown)
Responsible Party: Sponsor-Investigator, Bernardino Clavo, MD, PhD, MD, PhD, Head of Research Unit, Dr. Negrin University Hospital
Organization: Dr. Negrin University Hospital (Other)
Other Study IDs: DrNegrinUH; 2022-203-1 (Other: Ethics Committee of Las Palmas)
Record Dates: First submitted 2022-06-03; First posted 2022-06-14 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Radiation Toxicity; Chemotherapeutic Toxicity; Chemotherapy-induced Peripheral Neuropathy; Delayed Wound Healing; Chronic Pain; Refractory Pain
Keywords: Chemotherapy-induced Peripheral Neuropathy; Radiation-induced toxicity; Cancer-treatment side effects; Delayed wound healing; Chronic pain; Health-related quality of life; Anxiety and Depression; Ozone therapy; Refractory pain
MeSH Terms: conditions — Radiation Injuries; Chronic Pain; Pain, Intractable; Anxiety Disorders; Depression

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 28 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Ozone group: Patients treated with ozone as adjuvant palliative therapy. The procedure of ozone administration, dosage, frequency, and duration of ozone treatment will depend on the treated symptom and clinical evolution. Usually planned 40 sessions.
  Interventions: Other: Ozone therapy

INTERVENTIONS:
Other: Ozone therapy — Systemic and/or local ozone administration. Dosage, frequency, and duration of ozone treatment will depend on the treated symptom and clinical evolution. Usually planned 40 sessions.

SUMMARY:
The main objective of this study is to analyze the impact on the health-related quality of life of patients with refractory symptoms, who have been referred to the HUGCDN Chronic Pain Unit for adjuvant palliative treatment with ozone therapy between June-2022 and December-2025

DETAILED DESCRIPTION:
Chronic Pain Unit in the absence or failure of standard treatment, or when the standard treatment is associated with high morbidity or high risk. Frequently, these patients present alterations in self-perceived health-related quality of life (HRQoL), anxiety, depression, and other symptoms. This study aims to evaluate in these patients the effect of adjuvant symptomatic/palliative ozone therapy on the HRQoL and the potential changes from baseline on several parameters after treatment.

MAIN OBJECTIVES: To evaluate in these patients: 1) the clinical effect on the HRQOL of adding ozone to the standard treatment.

SECONDARY OBJECTIVES: To evaluate in these patients changes from baseline on 2) anxiety and depression, 3) pain (if applicable), 4) grade of toxicity (if applicable), 5) requirements of invasive procedures for symptom management, 6) evolution of main symptoms, 7) evolution of oxidative stress and inflammation (if systemic ozone therapy).

METHODOLOGY: Prospective and observational study of patients referred to our Chronic Pain Unit for symptomatic/palliative treatment with ozone therapy between 2022 and 2025.

MAIN VARIABLE: 1) HRQoL through the EQ-5D-5L questionnaire

SECONDARY VARIABLE: 2) anxiety and depression through the hospital anxiety/depression (HAD) questionnaire, 3) Pain through the visual analog scale (VAS), 4) grade of toxicity in cancer patients through the CTCAE v5.0 scale, 5) the number of invasive procedures required for symptom management, 6) self -reported percentage of symptom improvement, 7) biochemical parameters of oxidative stress and inflammation.

Assessments at weeks: 0 (baseline), 16 (end of O3/O2 treatment, objective), 28 (12 weeks after the end of ozone), and 40 (24 weeks after the end of ozone, control) Length of treatment: as required; initially, planned 16 weeks. Follow-up: 24 weeks after finishing O3/O2 treatment. Planned length of the clinical trial: 49 months.

ELIGIBILITY:
Inclusion Criteria:

1. Adults > = 18 years old.
2. Patients submitted to the Chronic Pain Unit of the Hospital Universitario de Gran Canaria Dr. Negrín for symptomatic/palliative treatment with ozone therapy because conventional treatment does not exist, it has been unsuccessful, or it is associated with high risk or high morbidity.
3. After evaluation of symptoms and patients, it exists a potential benefit of adding ozone treatment to the current treatment.
4. Patients have no contraindications for ozone treatment.
5. Patients have signed and dated the informed consent for the compassionated ozone treatment and the specific informed consent for this study

Exclusion Criteria:

1. Age < 18 years old.
2. Psychiatric illness or social situations that would limit compliance with study requirements.
3. Those who are incapable to fill in the scales used to measure variables.
4. Hemodynamically or clinically unstable patients or uncontrolled severe illness.
5. Uncontrolled cancer disease requiring chemotherapy treatment.
6. Life expectancy < 6 months
7. Contraindication or disability or to attend scheduled treatments.
8. Known allergy to ozone.
9. Pregnancy at the time of enrollment (for systemic ozone therapy). 10 Hemochromatosis (for systemic ozone therapy).

11. Known significant glucose-6-phosphate dehydrogenase deficiency (favism, acute hemolytic anemia) (for systemic ozone therapy).

12. Patients who do not meet all the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients submitted to the Chronic Pain Unit of the Hospital Universitario de Gran Canaria Dr. Negrín for symptomatic/palliative treatment with ozone therapy because standard treatment does not exist, it has been unsuccessful, or it is associated with high risk or high morbidity.
Sampling Method: Non-Probability Sample
Enrollment: 105 (Estimated)
Dates: Start 2022-06-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in the health-related quality of life by the "5-level, 5-dimension EuroQol" (EQ-5D-5L) questionnaire (at the end of ozone therapy) | 16 weeks
  Self-reported evaluation of: a) 5 physical and emotional items scored in five levels, from 1 (best: I have no problem) to 5 (worst: I have extreme problem or I am unable to…) and b) additional self-assessment of health by a visual analogue scale (0 = worst health patient can imagine, 100 = best health patient can imagine)

SECONDARY OUTCOMES:
Change from Baseline in Levels of anxiety and depression according to the hospital anxiety/depression scale (at the end of ozone therapy) | 16 weeks
  HAD scale is a self-administered questionnaire which assesses 14 items pertaining to symptoms of anxiety (seven) and depression (seven) experienced by patients. Each item is scored from 0 (better, no alteration) to 3 (worse level of alteration). For each symptom, overall score is from 0 (better, no anxiety or depression) to 21 (worse, very severe anxiety or depression).
Change from Baseline in pain score according to the visual analog scale (VAS) (at the end of ozone therapy) | 16 weeks
  Self-reported evaluation of the severity of pain according to the VAS, scored from 0 ("No pain") to 10 ("Pain as bad as you can imagine")
Change from Baseline in the grade of toxicity secondary to cancer-treatment (if applicable) according to the CTCAE v5.0 scale (at the end of ozone therapy) | 16 weeks
  Grade of toxicity secondary to cancer-treatment according to the CTCAE v5.0 (Common Terminology Criteria for Adverse Events from the National Cancer Institute) scale. Each toxicity is usually scored from 0 (asymptomatic or mild symptoms) to 5 (death).
Changes from Baseline in requirements of invasive procedures (surgery, blood transfusions, and therapeutic endoscopic procedures) required for symptom management (at the end of ozone therapy) | 16 weeks
  Number of invasive procedures (surgery, blood transfusions, and therapeutic endoscopic procedures) required for symptom management.
Changes from Baseline in the main symptoms (at the end of ozone therapy) | 16 weeks
  Self -reported percentage of symptom improvement from Baseline
Changes from Baseline in biochemical parameters of oxidative stress (if systemic ozone therapy) (at the end of ozone therapy). | 16 weeks
  Serum levels of biochemical parameters of oxidative stress
Changes from Baseline in biochemical parameters of inflammation (if systemic ozone therapy) (at the end of of ozone therapy). | 16 weeks
  Serum levels of pro-inflammatory cytokines
Change from Baseline in the health-related quality of life by the "5-level, 5-dimension EuroQol" (EQ-5D-5L) questionnaire. | 28 weeks
  Self-reported evaluation of: a) 5 physical and emotional items scored in five levels, from 1 (best: I have no problem) to 5 (worst: I have extreme problem or I am unable to…) and b) additional self-assessment of health by a visual analogue scale (0 = worst health patient can imagine, 100 = best health patient can imagine)
Change from Baseline in Levels of anxiety and depression according to the hospital anxiety/depression scale. | 28 weeks
  HAD scale is a self-administered questionnaire which assesses 14 items pertaining to symptoms of anxiety (seven) and depression (seven) experienced by patients. Each item is scored from 0 (better, no alteration) to 3 (worse level of alteration). For each symptom, overall score is from 0 (better, no anxiety or depression) to 21 (worse, very severe anxiety or depression).
Change from Baseline in pain score according to the visual analog scale (VAS). | 28 weeks
  Self-reported evaluation of the severity of pain according to the VAS, scored from 0 ("No pain") to 10 ("Pain as bad as you can imagine")
Change from Baseline in the grade of toxicity secondary to cancer-treatment (if applicable) according to the CTCAE v5.0 scale. | 28 weeks
  Grade of toxicity secondary to cancer-treatment according to the CTCAE v5.0 (Common Terminology Criteria for Adverse Events from the National Cancer Institute) scale. Each toxicity is usually scored from 0 (asymptomatic or mild symptoms) to 5 (death).
Changes from Baseline in requirements of invasive procedures (surgery, blood transfusions, and therapeutic endoscopic procedures) required for symptom management. | 28 weeks
  Number of invasive procedures ((surgery, blood transfusions, and therapeutic endoscopic procedures) required for symptom management.
Changes from Baseline in the main symptoms. | 28 weeks
  Self -reported percentage of symptom improvement from Baseline
Changes from Baseline in biochemical parameters of oxidative stress (if systemic ozone therapy). | 28 weeks
  Serum levels of biochemical parameters of oxidative stress
Changes from Baseline in biochemical parameters of inflammation (if systemic ozone therapy). | 28 weeks
  Serum levels of pro-inflammatory cytokines
Change from Baseline in the health-related quality of life by the "5-level, 5-dimension EuroQol" (EQ-5D-5L) questionnaire. | 40 weeks
  Self-reported evaluation of: a) 5 physical and emotional items scored in five levels, from 1 (best: I have no problem) to 5 (worst: I have extreme problem or I am unable to…) and b) additional self-assessment of health by a visual analogue scale (0 = worst health patient can imagine, 100 = best health patient can imagine)
Change from Baseline in Levels of anxiety and depression according to the hospital anxiety/depression scale. | 40 weeks
  HAD scale is a self-administered questionnaire which assesses 14 items pertaining to symptoms of anxiety (seven) and depression (seven) experienced by patients. Each item is scored from 0 (better, no alteration) to 3 (worse level of alteration). For each symptom, overall score is from 0 (better, no anxiety or depression) to 21 (worse, very severe anxiety or depression).
Change from Baseline in pain score according to the visual analog scale (VAS). | 40 weeks
  Self-reported evaluation of the severity of pain according to the VAS, scored from 0 ("No pain") to 10 ("Pain as bad as you can imagine")
Change from Baseline in the grade of toxicity secondary to cancer-treatment (if applicable) according to the CTCAE v5.0 scale. | 40 weeks
  Grade of toxicity secondary to cancer-treatment according to the CTCAE v5.0 (Common Terminology Criteria for Adverse Events from the National Cancer Institute) scale. Each toxicity is usually scored from 0 (asymptomatic or mild symptoms) to 5 (death).
Changes from Baseline in requirements of invasive procedures (surgery, blood transfusions, and therapeutic endoscopic procedures) required for symptom management. | 40 weeks
  Number of invasive procedures (surgery, blood transfusions, and therapeutic endoscopic procedures) required for symptom management.
Changes from Baseline in the main symptoms. | 40 weeks
  Self -reported percentage of symptom improvement from Baseline
Changes from Baseline in biochemical parameters of oxidative stress (if systemic ozone therapy). | 40 weeks
  Serum levels of biochemical parameters of oxidative stress
Changes from Baseline in biochemical parameters of inflammation (if systemic ozone therapy). | 40 weeks
  Serum levels of pro-inflammatory cytokines

CONTACTS AND LOCATIONS:
Overall Officials: Bernardino Clavo, MD, PhyD, Study Chair — Dr. Negrín University Hospital, Las Palmas, Spain; Pedro G Serrano-Aguilar, MD, PhyD, Study Director — Servicio de Evaluación. Servicio Canario de Salud. Spain; Bernardino Clavo, MD, PhyD, Principal Investigator — Dr. Negrín University Hospital, Las Palmas, Spain; Miguel A Caramés-Álvarez, MD, Principal Investigator — Dr. Negrín University Hospital, Las Palmas, Spain
Locations (1):
- Dr. Negrín University Hospital, Las Palmas, Las Palmas, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Clavo B, Martinez-Sanchez G, Rodriguez-Esparragon F, Rodriguez-Abreu D, Galvan S, Aguiar-Bujanda D, Diaz-Garrido JA, Canas S, Torres-Mata LB, Fabelo H, Tellez T, Santana-Rodriguez N, Fernandez-Perez L, Marrero-Callico G. Modulation by Ozone Therapy of Oxidative Stress in Chemotherapy-Induced Peripheral Neuropathy: The Background for a Randomized Clinical Trial. Int J Mol Sci. 2021 Mar 10;22(6):2802. doi: 10.3390/ijms22062802. PMID 33802143
- [Background] Clavo B, Navarro M, Federico M, Borrelli E, Jorge IJ, Ribeiro I, Rodriguez-Melcon JI, Carames MA, Santana-Rodriguez N, Rodriguez-Esparragon F. Long-Term Results with Adjuvant Ozone Therapy in the Management of Chronic Pelvic Pain Secondary to Cancer Treatment. Pain Med. 2021 Sep 8;22(9):2138-2141. doi: 10.1093/pm/pnaa459. No abstract available. PMID 33738491
- [Background] Clavo B, Navarro M, Federico M, Borrelli E, Jorge IJ, Ribeiro I, Rodriguez-Melcon JI, Carames MA, Santana-Rodriguez N, Rodriguez-Esparragon F. Ozone Therapy in Refractory Pelvic Pain Syndromes Secondary to Cancer Treatment: A New Approach Warranting Exploration. J Palliat Med. 2021 Jan;24(1):97-102. doi: 10.1089/jpm.2019.0597. Epub 2020 May 5. PMID 32379556
- [Background] Clavo B, Rodriguez-Esparragon F, Rodriguez-Abreu D, Martinez-Sanchez G, Llontop P, Aguiar-Bujanda D, Fernandez-Perez L, Santana-Rodriguez N. Modulation of Oxidative Stress by Ozone Therapy in the Prevention and Treatment of Chemotherapy-Induced Toxicity: Review and Prospects. Antioxidants (Basel). 2019 Nov 26;8(12):588. doi: 10.3390/antiox8120588. PMID 31779159
- [Background] Clavo B, Santana-Rodriguez N, Llontop P, Gutierrez D, Suarez G, Lopez L, Rovira G, Martinez-Sanchez G, Gonzalez E, Jorge IJ, Perera C, Blanco J, Rodriguez-Esparragon F. Ozone Therapy as Adjuvant for Cancer Treatment: Is Further Research Warranted? Evid Based Complement Alternat Med. 2018 Sep 9;2018:7931849. doi: 10.1155/2018/7931849. eCollection 2018. PMID 30271455
- [Background] Clavo B, Santana-Rodriguez N, Llontop P, Gutierrez D, Ceballos D, Mendez C, Rovira G, Suarez G, Rey-Baltar D, Garcia-Cabrera L, Martinez-Sanchez G, Fiuza D. Ozone Therapy in the Management of Persistent Radiation-Induced Rectal Bleeding in Prostate Cancer Patients. Evid Based Complement Alternat Med. 2015;2015:480369. doi: 10.1155/2015/480369. Epub 2015 Aug 18. PMID 26357522
- [Background] Clavo B, Santana-Rodriguez N, Gutierrez D, Lopez JC, Suarez G, Lopez L, Robaina F, Bocci V. Long-term improvement in refractory headache following ozone therapy. J Altern Complement Med. 2013 May;19(5):453-8. doi: 10.1089/acm.2012.0273. Epub 2012 Dec 7. PMID 23215625
- [Background] Clavo B, Ceballos D, Gutierrez D, Rovira G, Suarez G, Lopez L, Pinar B, Cabezon A, Morales V, Oliva E, Fiuza D, Santana-Rodriguez N. Long-term control of refractory hemorrhagic radiation proctitis with ozone therapy. J Pain Symptom Manage. 2013 Jul;46(1):106-12. doi: 10.1016/j.jpainsymman.2012.06.017. Epub 2012 Oct 26. PMID 23102757
- [Background] Clavo B, Santana-Rodriguez N, Lopez-Silva SM, Dominguez E, Mori M, Gutierrez D, Hernandez MA, Robaina F. Persistent PORT-A-CATH(R)-related fistula and fibrosis in a breast cancer patient successfully treated with local ozone application. J Pain Symptom Manage. 2012 Feb;43(2):e3-6. doi: 10.1016/j.jpainsymman.2011.09.002. No abstract available. PMID 22248793
- [Background] Clavo B, Suarez G, Aguilar Y, Gutierrez D, Ponce P, Cubero A, Robaina F, Carreras JL. Brain ischemia and hypometabolism treated by ozone therapy. Forsch Komplementmed. 2011;18(5):283-7. doi: 10.1159/000333795. Epub 2011 Oct 13. PMID 22105041
- [Background] Clavo B, Gutierrez D, Martin D, Suarez G, Hernandez MA, Robaina F. Intravesical ozone therapy for progressive radiation-induced hematuria. J Altern Complement Med. 2005 Jun;11(3):539-41. doi: 10.1089/acm.2005.11.539. PMID 15992242